CLINICAL TRIAL: NCT04658355
Title: Effect of Chlorhexidine Gluconate Versus Povidone-iodine on the Vaginal Microbiome as Vaginal Operative Preparation During Gynecologic Surgeries
Brief Title: Chlorhexidine Gluconate Versus Povidone-iodine
Acronym: CHDvPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Gabriella Smith, Resident Physician, University of Arizona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008991024
Record Dates: First submitted 2020-09-23; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Vaginal Flora Imbalance
MeSH Terms: interventions — chlorhexidine gluconate; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Chlorhexidine Gluconate vs Povidone-iodine group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone-Iodine (Active Comparator): Povidone-iodine to be used as the cleansing solution in this arm of patients for surgical vaginal preparation.
  Interventions: Other: Povidone-iodine
- Chlorhexidine Gluconate (Experimental): Chlorhexidine gluconate to be used as the cleansing solution in this arm of patients for surgical vaginal preparation.
  Interventions: Other: Chlorhexidine Gluconate

INTERVENTIONS:
Other: Chlorhexidine Gluconate — 4% Chlorhexidine Gluconate vaginal cleansing solution as a surgical preparation.
  Arms: Chlorhexidine Gluconate
Other: Povidone-iodine — 10% povidone-iodine vaginal cleansing solution as a surgical preparation.
  Arms: Povidone-Iodine

SUMMARY:
A hysterectomy, or removal of the uterus, is a common surgery performed for a variety of reasons. During this surgery, to prevent infection, the vagina is thoroughly prepped with a cleansing solution, most commonly chlorhexidine gluconate or povidone-iodine. While studies have shown that chlorhexidine gluconate is better at killing bacteria people have raised concerns on how it affects the vaginal tissue. It is important to study these effects the cleansing solution surgeons use for this surgery can not only prevent infection but not cause harmful side effects.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of different vaginal operative preparations on the vaginal tissue and microbiome. Our primary working hypothesis is that chlorhexidine prep is more deleterious to vaginal tissue than povidone-iodine preparations.

Hypothesis 1: chlorhexidine gluconate is more disruptive to the vaginal microbiome than povidone-iodine Hypothesis 2: chlorhexidine gluconate leads to more vaginal atrophy than povidone-iodine

ELIGIBILITY:
* Inclusion Criteria:

  1. Females
  2. all races and ethnicities
  3. English-speaking
  4. pre-menoupausal
  5. undergoing gynecologic surgeries requiring vaginal operative preparation at Banner University Medical Center - Phoenix.

Exclusion Criteria:

1. Patients with dx of vaginitis or vulvovaginal atrophy at time of surgery
2. Patients with an allergy to povidone-iodine and/or Chlorhexidine Gluconate
3. Individuals with any skin conditions, as determined by the physician, which could interfere with the conduct of the study or increase the risks to the test subject including any open or healing cuts/incisions, abrasions, or broken skin in the testing area as determined by the physician
4. Currently menstruating
5. Be using or have used antibiotics, antifungals, topical steroids or antiviral (oral or topical in the testing areas) less than 12 weeks prior to visit
6. Have a history of or current, self-reported genital herpes
7. Have current or in the past 6 weeks, conditions such as

   1. Vaginal infection/bacterial vaginosis/yeast infection or sexually transmitted infection (Chlamydia, Gonorrhea or Trichomonas)/Hepatitis/HIV
   2. Vulvar infection
   3. Urinary tract infection
8. Sexual intercourse less than 48 hours prior to the visit
9. Current treatment for any skin conditions on the testing area

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of patient-reported vaginal and urinary symptoms after treatment with chlorhexidine gluconate or povidone-iodine vaginal cleansing solution | From date of surgery to 24 hours post-operative
  To compare the frequency of patient-reported vaginal and urinary symptoms after treatment with chlorhexidine gluconate or povidone-iodine vaginal cleansing solution utilizing questionnaires.

SECONDARY OUTCOMES:
Relative abundances of vaginal microbiota species | From date of surgery to 3-6 weeks postoperative
  To measure the change in relative abundances of vaginal microbiota species after treatment with chlorhexidine gluconate or a povidone-iodine vaginal cleansing solution. Vaginal microbiota species include but not limited to health-associated Lactobacillus spp., bacterial-vaginosis associated anaerobes (Gardnerella, Prevotella, Sneathia, Atopobium, Megasphaera, Parvimonas, Mobiluncus and others), pathobionts (Streptococcus, Escherichia), and other bacterial taxa present in the collected vaginal swabs using 16S rRNA sequencing

OTHER OUTCOMES:
Change in level of genital cytokines and chemokines | From date of surgery to 3-6 weeks post-operative
  To measure the change in levels of genital cytokines and chemokines (IL-1alpha, IL-1beta, IL-8, MIP-1beta, MIP-3alpha, RANTES, TNFalpha) in the collected cervicovaginal lavages using multiplex cytometric bead arrays after treatment with chlorhexidine gluconate or a povidone-iodine vaginal cleansing solution. The cytokine levels will be used to determine the genital inflammatory score by using a previously described genital inflammation scoring system. Patients will be assigned one point for each mediator when the level was in the upper quartile
Change in vaginal pH level | From date of surgery to 3-6weeks post-operative
  To measure the change vaginal pH after treatment with chlorhexidine gluconate or a povidone-iodine vaginal cleansing solution.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Foley, MD, Study Chair — Banner University Medical Center - Phoenix/ University of Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Niaimi A, Rice LW, Shitanshu U, Garvens B, Fitzgerald M, Zerbel S, Safdar N. Safety and tolerability of chlorhexidine gluconate (2%) as a vaginal operative preparation in patients undergoing gynecologic surgery. Am J Infect Control. 2016 Sep 1;44(9):996-8. doi: 10.1016/j.ajic.2016.02.036. Epub 2016 May 24. PMID 27234011
- [Background] Amstey MS, Jones AP. Preparation of the vagina for surgery. A comparison of povidone-iodine and saline solution. JAMA. 1981 Feb 27;245(8):839-41. PMID 7463676
- [Background] Aronson JK. Antiseptic drugs and disinfectants. In: Side effects of drugs annual. Vol 35. Elsevier Science & Technology; 2014:435-445. https://www.sciencedirect.com/science/article/pii/B9780444626356.000243. 10.1016/B978-0-444-62635-6.00024-3.
- [Background] American College of Obstetricians and Gynecologists Women's Health Care Physicians; Committee on Gynecologic Practice. Committee Opinion No. 571: Solutions for surgical preparation of the vagina. Obstet Gynecol. 2013 Sep;122(3):718-20. doi: 10.1097/01.AOG.0000433982.36184.95. PMID 23963423
- [Background] Costin GE, Raabe HA, Priston R, Evans E, Curren RD. Vaginal irritation models: the current status of available alternative and in vitro tests. Altern Lab Anim. 2011 Sep;39(4):317-37. doi: 10.1177/026119291103900403. PMID 21942546
- [Background] Culligan PJ, Kubik K, Murphy M, Blackwell L, Snyder J. A randomized trial that compared povidone iodine and chlorhexidine as antiseptics for vaginal hysterectomy. Am J Obstet Gynecol. 2005 Feb;192(2):422-5. doi: 10.1016/j.ajog.2004.08.010. PMID 15695981
- [Background] Fleischer W, Reimer K. Povidone-iodine in antisepsis--state of the art. Dermatology. 1997;195 Suppl 2:3-9. doi: 10.1159/000246022. PMID 9403248
- [Background] Lewis LA, Lathi RB, Crochet P, Nezhat C. Preoperative vaginal preparation with baby shampoo compared with povidone-iodine before gynecologic procedures. J Minim Invasive Gynecol. 2007 Nov-Dec;14(6):736-9. doi: 10.1016/j.jmig.2007.05.010. PMID 17980335
- [Background] Mac Bride MB, Rhodes DJ, Shuster LT. Vulvovaginal atrophy. Mayo Clin Proc. 2010 Jan;85(1):87-94. doi: 10.4065/mcp.2009.0413. PMID 20042564
- [Background] Mahoney JB, Chernesky MA. Institutional infection control and prevention. Manual of clinical microbiology. 1999:108-190.
- [Background] Rastogi S, Glaser L, Friedman J, Carter IV, Milad MP. Tolerance of chlorhexidine gluconate vaginal cleansing solution: A randomized controlled trial. Journal of Gynecologic Surgery. 2019. doi: 10.1089/gyn.2019.0066.
- [Background] US National Library of Medicine.4% chlorhexidine gluconate skin cleansing kit; US food and drug administration (FDA) approved product information. DailyMed Web site. https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=65f87900-8d23-4fb3-be44-1d116aedac78. Updated 2015.
- [Background] Vorherr H, Vorherr UF, Mehta P, Ulrich JA, Messer RH. Antimicrobial effect of chlorhexidine and povidone-iodine on vaginal bacteria. J Infect. 1984 May;8(3):195-9. doi: 10.1016/s0163-4453(84)93811-8. PMID 6736662
- [Background] Wilkinson EM, Laniewski P, Herbst-Kralovetz MM, Brotman RM. Personal and Clinical Vaginal Lubricants: Impact on Local Vaginal Microenvironment and Implications for Epithelial Cell Host Response and Barrier Function. J Infect Dis. 2019 Nov 6;220(12):2009-2018. doi: 10.1093/infdis/jiz412. PMID 31539059